CLINICAL TRIAL: NCT00323973
Title: A Randomized Double-blind Placebo Force-titration Controlled Study With Bisoprolol in Patients With Chronic Heart Failure Secondary to Chagas´ Cardiomyopathy.
Brief Title: Chagas Cardiomyopathy Bisoprolol Intervention Study: Charity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Victor Castillo, Executive Director, Fundación Cardiovascular de Colombia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: fcv059
Record Dates: First submitted 2006-05-05; First posted 2006-05-10 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Chagas Cardiomyopathy; Chronic Heart Failure
Keywords: Chagas, Heart failure, Cardiomiopathy
MeSH Terms: conditions — Chagas Cardiomyopathy; Heart Failure | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bisoprolol
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — 10 mg qd
  Other Names: Bisoprex

SUMMARY:
Chagas disease (CD) is the major cause of disability secondary to tropical diseases in young adults from Latin America. In this region 20 million people are currently infected by T. cruzi, the etiologic agent for CD. In Colombia, 18 percent of the population live in CD endemic areas, 900,000 people are infected and over three million are at high risk of being infected. Heart failure due to Chagas cardiomyopathy (CCM) is the main clinical form of CD in Colombia. However, the incidence of CCM among T. cruzi infected people is unknown and the mechanisms that lead from infection to CCM are uncertain. Besides the poor prognosis of CHF due to Chagas disease, it is important to estimate the risk of complications and death in patient infected with T. cruzi Unfortunately, few clinical studies have addressed this issue. Most T. cruzi infected patients have mild or no clinical disease, however, the percentage of infected people that will develop detectable cardiac abnormalities is approximately 30 to 40 percent, but only 20 percent of them will develop symptomatic cardiac involvement. Like CHF from other causes, CHF due to CD responds to digital, diuretics and vasodilators therapy. Also, some studies have shown that angiotensin-converting enzyme (ACE) inhibitors improve survival in patients with moderate to severe CHF due to CD. Increased sympathetic drive results in an increased risk of cardiac arrhythmia and sudden death. Beta-adrenoreceptor antagonism seems to protect against the deleterious effects of chronic sympathetic stimulation. The effects of the selective beta-adrenergic receptor blocker Bisoprolol on cardiovascular mortality, hospital readmission due to progressive heart failure and functional status in patients with CHF secondary to CCM has not been explored to-date. To evaluate the benefit of Bisoprolol in CHF due to CCM, a cohort of T. cruzi seropositive patients will be selected from several institutions in Colombia. Patients will be classified according to a modified version of the Panamerican Health Organization recommendations for patients with CCM. Overall one year mortality in patients with CHF due to Chagas disease has been reported as 34 percent. However, one year mortality is only 3 percent in patients in NYHA functional class II, 27 percent in those in NYHA functional class III, and 62 percent among those in functional class IV (22). The sample size has been calculated assuming an event rate of 40 percent in two years in the placebo group, and using a 95 percent confidence level and power of 80 percent, we will need to recruit 250 patients per treatment arm to detect a reduction of 30 percent in the risk of the primary outcome. The event rate we have used to estimate sample size is similar to the expected two-year mortality in patients with CHF due to Chagas disease in NYHA functional class II. Therefore, the estimated sample size should be enough to measure significant changes in the composite primary outcome (death, HF hospitalizations, SMVT, SCD). The recruitment process will follow guidelines set out by the FCV Ethics Committee. Most participants will be recruited from the Chagas disease and the Heart Failure clinics located in Bucaramanga, Bogotá and Cucuta. During the pretreatment period an initial evaluation visit will be scheduled in which participants will sign consent forms, baseline measurements and tests will be conducted at the FCV including blood pressure measurements obtained with patients in the sitting and standing positions. Laboratory test such as twelve-lead ECG will be recorded in each patient. Left ventricular ejection fraction at rest will be determined by 2D echocardiography, using a modified Simpsons rule to calculate LV volumes. Quality of life questionnaire will be performed two weeks apart during baseline examination using the Minnesota living with heart failure questionnaire. Minimum of two 6-minutes corridor walk test once a week over a two-week period will be performed to measure the functional class. During the treatment period patients will be randomly assigned to receive double-blind Bisoprolol or placebo, initially taking a total daily dose of 2.5 mgrs qd. The dose will be increased every two weeks to 5 up to 7.5 and 10 mgrs qd (maximum maintenance dose). Follow-up assessment will include clinical check-up, and blood collection for future measurements of inflammatory reactants and markers. Quality of life measurements will be obtained at six months. Following the descriptive analysis we will compare the patient survival and hospitalization rates using Kaplan-Meier estimates and survival graphs. Cox regression will be used for the multivariate analysis of time to death and time to hospitalization. This analysis will allow us to explore the pattern of changes in patients with chronic heart failure due to Chagas disease such as the effect of beta-blockers in this special type of cardiomyopathy.

DETAILED DESCRIPTION:
BACKGROUND

Chagas disease (CD) is a permanent threat for almost a quarter of the population of Latin America. Although the disease has been described in almost all Central and South America, clinical presentation and epidemiological characteristics are highly variable among the different endemic zones (1,2). A wide range of prevalence rates has also been reported suggesting local differences in transmission of the disease as well as differences in vectors and reservoirs (3). Chagas cardiomyopathy (CCM) represents a serious public health problem in most Latin American countries, and the most recent statistics provided by the World Health Organization indicate that 100 million persons are exposed to the disease and approximately 20 million are currently infected (4). Interestingly, in addition to the natural infection foci, an increase in the transmission associated with blood transfusions has also been noticed. These statistics are considered an underestimation of the real rates of infection, most likely due to lack of reports from highly endemic retired rural communities. In countries in which the disease is endemic such as Colombia, Venezuela and Brazil, the overall prevalence of infection averages 10 percent. However, in highly endemic rural areas rates have ranged from 25 to 75 percent (5). Prevalence of infection varies widely even between cities and provinces within the same country because of variations in climate, housing condition, public health measures, and urbanization. The actual prevalence of clinical Chagas disease and the number of case fatalities are largely unknown, mainly because case reporting is virtually nonexistent in many areas in which CD is highly endemic. Congestive heart failure (CHF) is a late manifestation of CD that results from structural abnormalities and extensive and irreversible damage to the myocardium. Heart failure in T. cruzi infected patients usually occurs after age 40 and follows AV block or ventricular aneurysm. However, when CHF develops in patients less than 30 years old it is frequently associated with a more aggressive myocarditis and an extremely poor prognosis (1). The mortality attributable to CD is related to the severity of the underlying heart disease. Very high mortality is often found in patients with congestive heart failure (2), however, mortality in asymptomatic seropositive patients varies greatly between geographic regions, suggesting that other factors may influence the severity and progression rate of cardiac disease. It is believed that cardiac damage in CD progresses slowly but steadily over decades, from subclinical myocarditis to mild segmental abnormalities with conduction defects, to severe ventricular structural abnormalities, and finally to overt congestive heart failure and sudden cardiac death.

Besides the poor prognosis of CHF due to Chagas disease, it is important to estimate the risk of complications and death in patient infected with T. cruzi. Unfortunately, few clinical studies have addressed this issue. Most T. cruzi infected patients have mild or no clinical disease, however, the percentage of infected people that will develop detectable cardiac abnormalities is approximately 30 to 40 percent (3), but only 20 percent of them will develop symptomatic cardiac involvement (6). Like CHF from other causes, CHF due to CD responds to digital, diuretics and vasodilators therapy (7). Additionally, some studies have shown that angiotensin converting enzyme (ACE) inhibitors improve survival in patients with moderate to severe CHF due to CD (8). In spite of its benefits on patients with non Chagas disease CHF, there is considerable uncertainty about the potential role of ACE inhibitors in patients with CHF due to Chagas disease. Captopril, and ACE inhibitors, has been shown to reduce neurohormonal activation and non lethal arrhythmias in a small number of patients with Chagas heart failure (8,9). Another intervention currently included in the management of CHF patients is the use of b blockers. Observational studies (10) as well as clinical trials (11,12) have shown that b-blockers reduce morbidity and mortality in CHF patients. The effects of b-blockers on CHF patients are being studied in large scale clinical trials (13-19). Apparently, the cardiac sympathetic hyperstimulation that initially helps to preserve ventricular function in CHF patients, later on, results in an increased risk of cardiac arrhythmia and sudden death (20) b-adrenoreceptor antagonism seems to protect against the deleterious effects of chronic sympathetic stimulation (21). Moreover, b-blockers reduce heart rate, improve myocardial energetic balance and lead to a less negative force-frequency relationship. These effects contribute to the benefits of b-blocker therapy in CHF patients. Clinical studies with Carvedilol, a a1 and non selective b-blocker, further support the beneficial effects of b-adrenoceptor antagonism (18,19,23,24). Results from the US CARVEDILOL and COPERNICUS trial, suggest that prognosis in CHF may partly depend on left ventricular dysfunction improvement as well as sympathetic activity reduction (18,23). However, additional data are needed to define more precisely the relationships between heart rate reduction, left ventricular function improvement and survival in CHF patients. In some studies like CIBIS II and MERIT HF, the beneficial effects of the selective b- blockers on morbidity and mortality were observed specially in patients functional class II and III. In COPERNICUS a multicentric placebo controlled clinical trial with Carvedilol, these effect was ascertained even in patients functional class IV (23), demonstrating that patients with CHF, independently of their functional class, should receive b-blocker therapy. Current guidelines for the management of CHF strongly recommend the use of beta-blockade in management of CHF. However, these benefits have not been proven in Chagas´ cardiomyopathy (25,26). Nevertheless, there are reasons to believe that beta-blockade will be beneficial for these patients.

First, patients with CHF due to CD have a raised end-diastolic pressure associated with a low systemic blood pressure, which lead to low transmyocardial pressure gradient and subendocardial ischemia. Therefore, reduction in myocardial oxygen demand due to beta-blockade could be expected to be beneficial in this situation, even in non ischemic CHF patients. Second the reduction in sudden cardiac deaths and serious ventricular arrhythmias suggest that an anti arrhythmic effect is an important component of beta-blockade. This anti-arrhythmic effect is explicable not only on an anti-ischemic basis but also by blockade of sympathetic activity, which is indeed increased in patients with Chagas cardiomyopathy. Third, prolonged activation of the sympathetic nervous system can accelerate the progression of heart failure, and the rate of progression can be substantially decreased using pharmacological agents that interfere with sympathetic activity in the heart and peripheral blood vessels. There is clear evidence of increased circulating beta-adrenergic antibodies in Chagas disease providing further theoretical support for the use of beta-adrenergic blockade in this group of patients.

Beta-blockers already proven to be beneficial in CHF patients are metoprolol, bisoprolol and carvedilol, drugs which have been tested in over 10.000 patients in more than 20 placebo-controlled clinical trials enrolling men and women with systolic dysfunction due to ischemia, hypertension and dilated idiopathic cardiomyopathy.

Bisoprolol is a beta-1 selective blocker with the highest selectivity for this receptor, in doses less than 10 mg it has very little or no effect on beta-2 receptors. Bisoprolol was first tested in CHF in the CIBIS I trial which enrolled 641 patients and showed improvement in functional class, less hospitalizations for heart failure and a trend to improved survival. The much larger randomized CIBIS II assigned 2647 patients with class III or IV HF and an LVEF lower than 40 percent to bisoprolol or placebo, the patients also received standard therapy with diuretics and ACE inhibitors. After an average follow-up of 1.4 years, the trial was prematurely stopped when the benefits were observed in the active treatment group: significant reduction in total all-cause mortality (11.8 versus 17.3 percent) that was independent of the severity or cause of HF. This benefit was primarily due to a reduction in SCD (3.6 versus 6.3 percent, p 0.001), with a non-significant trend toward fewer deaths from HF, significant 15 percent reduction in hospital admissions for any cause and a 30 percent reduction in admissions for HF (p 0.0001).

Considering all the beneficial effects beta-blockers in patients with mild to severe CHF due to ischemic and non ischemic disease, there is no data regarding its potential effects in patients with CHF due to Chagas disease. Based on the aforementioned we propose to develop a multi-center placebo controlled clinical trial to evaluate the effect of Bisoprolol in patients with CHF due to CD.

OBJECTIVES

Primary Objective:

To investigate the effect of the beta-blocker bisoprolol on survival and HF hospitalization rates, and other previously predefined outcomes in patients with Chagas cardiomyopathy and heart failure.

Secondary Objective:

To investigate the effect of the beta-blocker bisoprolol on quality of life, progression to heart block and need for electrical therapy (i.e. pacemaker, ICD, CRT).

OUTCOMES

Primary Outcomes:

The composite of the first occurrence of ANY of the following

* Cardiovascular death.
* Hospital admission caused by heart failure.
* Major adverse cardiovascular events: stroke, systemic embolism, resuscitated sudden death.
* Bradycardia requiring pacemaker implantation.
* Clinically significant sustained monomorphic ventricular tachycardia causing syncope: sustained ventricular tachycardia or ventricular fibrillation.

Secondary Outcomes:

* Non-cardiovascular death.
* Heart failure worsening or mortality related with CHF.
* New AV block.
* Need for Implantable cardioverter-defibrillator (ICD), Cardiac resynchronization Therapy (CRT) or Pacemaker therapy (PM).
* Perceived quality of life worsening.

HYPOTHESES

* Bisoprolol will reduce cardiovascular death in patients with Chagas cardiomyopathy with heart failure functional class NYHA II to IV.
* Bisoprolol is safe in patients without advanced heart block.
* Bisoprolol will significantly reduce hospitalization rates due to heart failure in patients with Chagas cardiomyopathy in functional class NYHA II to

STUDY DESIGN

CHARITY is a multicenter randomized prospective, double blind, placebo-controlled, forced-titration study in subjects with CHF secondary to CCM. Enrolled subjects will receive placebo or Bisoprolol in addition to standard therapy for chronic heart failure which includes an ACE-inhibitor and may include diuretics or other medication such as digitalis or nitrates for heart failure.

Patients included in CHARITY should be on stable doses of an ACE-inhibitor. Diuretics can be added to treatment as needed but patients must be on stable doses of each drug during four weeks prior to randomization.

500 subjects will be randomized in two arms; one will receive oral bisoprolol and the other placebo, during the duration of the study. Forced titration will start with the lowest oral dose of 2.5 mg qd and will be up-titrated in 2.5 mg increments every two weeks until the maximum tolerated dose is achieved or 10 mg qd is reached. In case of intolerance, dose will be reduced to the previously tolerated lower dose. Subjects not tolerating the lower dose of 2.5 qd will have a treatment interruption. The best tolerated dose will be continued for one month, then a security visit will re-asses tolerance. Thereafter patients will be controlled every three months until they complete the mean follow-up period of two years. Standard heart failure therapy with ACE-inhibitors, diuretics, digitalis and nitrates will be strongly reinforced in both parallel arms.

BLINDING

Patients and investigators will remain blinded during the trial. The treatment codes will remain blinded until the database is locked for final analysis.

PRETREATMENT CONSIDERATIONS

Baseline vital signs will be obtained with patients in the sitting and after 3 minutes in the standing position.

Twelve-lead ECGs will be recorded in each patient. Left ventricular ejection fraction at rest will be determined by echocardiography, using a modified Simpsons rule to calculate LV volumes.

Quality of life questionnaire will be administrated two weeks apart during baseline examination using a translated-validated version of the Minnesota living with heart failure questionnaire.

Minimum of two 6-minutes corridor walk test once a week over a 2-week period will be performed. The last value will be used if it is within 10 percent of the previous value.

FOLLOW-UP PERIOD

ECG tracings will be recorded during the security visit and at 1 and 2 years. Patients will be followed for two years after randomization. Repeat echocardiograms will be recorded at 1 and 2 years of follow-up along with HF Quality of-life questionnaire and six-minute walk tests.

Clinical measurements will be obtained every three months along with an assessment of treatment adherence and tolerance. Mortality and hospitalization events will be ascertained by telephonic interview and verified with hospital charts review, up to two years after randomization.

MONITORING COMMITTEES

Steering committee

The committee has the overall responsibility for producing and conducting a scientifically sound design and ensuring accurate reporting of the study. In that capacity, the Steering Committee must address and resolve scientific issues encountered during the study. This committee will meet at least twice a year. The main role of the Steering Committee is the development of the protocol and CRF and to ensure appropriate conduction of the trial. The steering committee is composed by the principal investigators and site investigators. The chairman of the steering committee is the principal investigator. The primary scientific publication reporting the study results is the responsibility of the Steering Committee.

CHARITY Operations Committee

The Operations Committee will consist of a select group of Steering Committee members chosen for their specific expertise and experience. This group will be responsible for ensuring that study execution and management are of the highest quality.

FCVRI Project Office

The FCVRI Project Office is located at the Instituto de Investigaciones-FCV in Bucaramanga, Santander, Colombia,is independent and its primary function is to facilitate and oversee the execution of the study. The FCV Project Office will keep the Operations Committee appraised of the progress and conduct of the trial and will provide ongoing administrative and methodological support to the Event Adjudication Committee and the DSMB

Data and Safety Monitoring Board (DSMB)

The DSMB will include at least 2 prominent cardiologists and a neurologist, as well as a statistician. Their mandate will be to provide on-going review of the safety of all the investigational treatments.

Adverse Events and Adjudication Committee

The Event Adjudication Committee is charged with the responsibility for validating all reported primary fatal and nonfatal outcomes and validating the classification of cause of death. The Event Adjudication process will be coordinated at the FCVRI Project Office in Bucaramanga. This committee, composed of experts in the field will review, in a blinded manner; all reported outcome events to provide consistency and validity in the assessment of outcomes. Their decisions will be based on blind clinical data provided and they will consider the impressions of the clinical investigator. Their decisions will be used in the final analysis. The AE Committee (AE-AC) is composed by clinical experts and one principal investigator, its responsibilities are to review and verify every AE, SAE and Adverse Drug Reactions (ADR) reported, and to supervise all relevant SAE information is complete. The AE-EC will validate all SAE in a blinded form and notify investigators, Independent Ethics Committees and regulation authorities of all SAE and clinically relevant AE. The AE-EC will also validate outcomes providing standard classifications and definitions and reviewing supporting information provided by investigators.

SELECTION AND WITHDRAWAL OF SUBJECTS

Inclusion Criteria

* Males or females aged 18 to 70 years.
* Heart failure symptoms NYHA functional class II to IV
* Left ventricular ejection fraction lower than 40 percent determined by bi-dimensional echocardiography using modified Simpsons rule for ventricular volumes.
* Subjects must be on standard and stable outpatient doses of ACEIs or angiotensin II receptor antagonist for at least four weeks.
* Subjects receiving diuretics must be on a stable dose for at least two weeks.
* Clinical Euvolemia:as evidenced by absence of rales, no pleural effusion or ascitis and no more than minimal peripheric edema.

Exclusion Criteria

* CHF due to ischemic heart disease, valvular disease or any other etiology different than CD.
* Severe aortic insufficiency
* Baseline advanced AV block defined as Mobitz type 2 or third degree AV block
* Serum creatinine greater than 2.5 mg/dl.
* Resting Heart rate less than 45 bpm
* Known malignancy and other severe disease which shorten life expectancy less than 6 months.
* Subjects with contraindications for beta-blockers: severe obstructive chronic pulmonary disease, asthma, severe pulmonary hypertension, type 1 diabetes mellitus or history of hypoglycemia.
* Suspected or confirmed chronic infectious disease including HIV and hepatitis B.
* History of active substance or alcohol abuse within the last year.
* Clinically significant psychiatric illness which can negatively affect the subject compliance and participation in the trial.
* Pregnancy or lactation.
* Organic disease or gastrointestinal surgery which can affect the oral absorption and pharmacodynamics of the medication under study.
* Enrollment and participation in other active treatment trial within the previous month.
* Failure to provide written informed consent.

Interruption of treatment

Trial treatment should be interrupted under the following conditions.

* The patient decides it is in his-her best interest.
* The investigator considers it is advisable or in the patients best interest.
* Intolerable adverse experience(s).
* Presence of life-threatening conditions despite adjustment of therapy.

If study treatment is interrupted, every effort should be made to reinstate treatment as soon as possible and medically acceptable. The re-initiation dose is determined at investigators discretion and the dose may be reduced or re-started at the last dose level. Patients with treatment interruption should continue on the protocols visit schedule and study procedures except drug dispensing.

TREATMENTS

The FCV Research Institute will supply ranurated 5 mg bisoprolol tablets and matched placebo needed for the whole duration of the trial. Study drug and placebo have been kindly provided by Merck Colombia.

EFFICACY ASSESSMENT

Efficacy assessments will be made at every visit during the trial following randomization. Information will be recorded in the supplied CRF formats dealing with clinical variables, Adverse Events (AE), Serious Adverse Events (SAE) and endpoints.

Each of the primary endpoints will be recorded on the SAE form and in the individual corresponding form for each endpoint.

Endpoint Definitions

Cardiovascular death: any death attributable to a cardiac or vascular cause occurring within two years after randomization.

Non-cardiovascular death: death from any cause excluding cardiovascular diseases occurring within two years after randomization..

Hospital admission-hospitalization caused by heart failure: admission in a hospital or clinic during at least 24 hours caused by heart failure worsening. It excludes procedures and hospitalization for procedures which have been scheduled and not due to worsening of the current heart failure condition since randomization.

Heart failure worsening: decline of at least one functional class as defined by the New York Heart Association occurring during any inter-visit period of three months needing inotropic support, IV diuretics, medication dose adjustments or additional drugs for compensation.

Perceived quality of life worsening: increase in the Minnesota living with heart failure test score of at least 10 points. The tests score ranges from 0 (best) to 100 (worst).

New AV block: appearance of any AV conduction disturbance including first, second and third degree AV block after randomization.

Bradycardia requiring pacemaker implantation: ventricular rates < 50 per minute due to any cause including sick-sinus syndrome and AV block, causing symptoms or disability and complying with current indications for permanent pacemaker implantation.

ICD: Implantable cardioverter-defibrillator indicated for the prevention and treatment of sudden death, ventricular tachycardia/ventricular fibrillation.

CRT: cardiac resynchronization therapy or biventricular pacing or ventricular bifocal pacing for the treatment of advanced heart failure.

PM: permanent pacemaker for the treatment of conduction disturbances. Clinically significant ventricular arrhythmias: sustained monomorphic ventricular tachycardia or ventricular fibrillation with symptoms caused by hemodynamic or perfusion alterations, circulatory collapse or syncope.

STATISTICAL METHODS

Descriptive statistical analysis will be composed with simple distribution of frequencies, calculation of proportions, means, their respective standard deviations and 95 percent confidence intervals. For effects of group comparison, t-test and Mann-Whitney tests will be used according to the dependent variable distribution. For categoric variables, the Chi-square test or the exact Fisher test will be applied as corresponding.

Patient survival and hospitalization rates will be described using Kaplan-Meijer estimates and survival graphs. Cox regression will be used for the multivariate analysis of time to death and time to hospitalization.

Formal efficacy interim analyses will take place one year after the recruitment phase.

Expected Results

Direct Results: Study results will help identify interventions potentially useful to prevent the progression from T. cruzi infection to CCM. This may significantly lessen the burden of CD in Colombian and other exposed populations. This will have a significant impact on the morbidity and mortality of the Colombian population, mainly in areas with high prevalence of seropositive subjects for T. cruzi such as Santander. The execution of this project will allow us to determine the effect of the b-blocker therapy on the CCM and the behavior of the autonomic nervous system on the mortality and morbidity of subjects infected by T. cruzi. The results of this study will also arise the need knowledge to suggest new therapeutic interventions for patients with CCM.

Indirect Results: This project will contribute to the consolidate the clinical research group of the Easter Cardiovascular Foundation as well the Chagas group that is already working at the same institution.

Strategy to be use for data transferring

According to recent trends in the field literature we will try to get the results of this project in one of the following clinical journals: Circulation, Journal of the American College of Cardiology, American Journal of Cardiology and another one in one of the following basic journals: Infection and Immunity, Transactions of the Royal Society of Tropical Medicine and Hygiene. The obtained results from this study will be presented at the Colombian Congress of Cardiology, the Colombian Congress of Intern Medicine and at least in one international meeting (Inter American Congress of Cardiology, Meeting of the American College of Cardiology or the Annual Meeting of the American Heart Association). This strategy will guarantee the communication, discussion and evaluation of the results by the international scientific community in this subject.

Experience of the Research Group and presentation of the research team.

The members of the research team belong to the Research Institute of the Fundación Cardiovascular del Oriente Colombiano (RIFCV) are physician from the medical staff of the FCV and from the Instituto Colombiano de Investigacion ICIB, one of the members of the VILANO group. The RIFCV is a well recognized research center, that has been promoted by COLCIENCIAS, and has received twice economical support. During the last tree years the RIFCV has been funded by COLCIENCIAS to make five research projects. Two of them, related to this subject, are being carried out right now. Moreover, the RIFCV has also been funded by the Ministry of Health for two projects. The RIFCV has also participated in more than ten projects funded by pharmaceutical companies.

The RIFCV is one of the institution that constitute the ICIB. Three of the researcher of this project, (CAM, LAC, JPC ) belong to the VILANOs group, which has been qualified by COLCIENCAS as a group class A. The research team is a multidisciplinary group constituted by physicians of several fields (Basic science, clinic and epidemiology) and includes one masters, tree cardiologist, one master student and two general physician. The high academic degree and the experience of the group allow to carry out high degree research with good quality. Tree of the members of the team has developing research in the autonomic aspects of CCM and one have been working in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 70 years.
* Heart failure symptoms NYHA functional class II to IV
* Left ventricular ejection fraction <40% determined by bi-dimensional echocardiography using modified Simpson's rule for ventricular volumes.
* Subjects must be on standard and stable outpatient doses of ACEIs or angiotensin II receptor antagonist for at least four weeks.
* Subjects receiving diuretics must be on a stable dose for at least two weeks.
* Clinical Euvolemia:as evidenced by absence of rales, no pleural effusion or ascitis and no more than minimal peripheric edema.

Exclusion Criteria:

* CHF due to ischemic heart disease, valvular disease or any other etiology different than CD.
* Severe aortic insufficiency
* Baseline advanced AV block defined as Mobitz type 2 or third degree AV block
* Serum creatinine >2.5 mg/dl.
* Resting Heart rate less < 45 bpm
* Known malignancy and other severe disease which shorten life expectancy < 6 months.
* Subjects with contraindications for beta-blockers: severe obstructive chronic pulmonary disease, asthma, severe pulmonary hypertension, type 1 diabetes mellitus or history of hypoglicemia.
* Suspected or confirmed chronic infectious disease including HIV and hepatitis B.
* History of active substance or alcohol abuse within the last year.
* Clinically significant psychiatric illness which can negatively affect the subject compliance and participation in the trial.
* Pregnancy or lactation.
* Organic disease or gastrointestinal surgery which can affect the oral absorption and pharmacodynamics of the medication under study.
* Enrollment and participation in other active treatment trial within the previous month.
* Failure to provide written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hospital admission caused by heart failure. | 2 years
Major adverse cardiovascular events: stroke, systemic embolism, resuscitated sudden death. | 2 years
Bradycardia requiring pacemaker implantation. | 2 years
Clinically significant sustained monomorphic ventricular tachycardia causing syncope: sustained ventricular tachycardia or ventricular fibrillation. | 2 years

SECONDARY OUTCOMES:
Non-cardiovascular death. | 2 years
Heart failure worsening or mortality related with CHF. | 2 years
New AV block. | 2 years
Need for Implantable cardioverter-defibrillator (ICD), Cardiac resynchronization Therapy (CRT) or Pacemaker therapy (PM). | 2 years
Perceived quality of life worsening. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Morillo, MD, FRCPC, Principal Investigator — Fundación Cardiovascular de Colombia
Locations (1):
- Fundación Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia